CLINICAL TRIAL: NCT05130008
Title: Implementing a Digitally-enabled Community Health Worker Intervention for Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jocelyn Carter, Physician- Scientist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018P002014; 1K23HL150287-01 (NIH)
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure，Congestive
Keywords: community health worker care; digital platform; remote monitoring; readmissions; clinical trial; heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor team will be blinded to the intervention assignments of participants. Due to the nature of the intervention, the participants, the investigator, and the care providers are unable to be blinded to the participant assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients identified by the MGH readmission database and the EHR as eligible for the study will be enrolled. Participants will be paired with a community health worker and oriented to the digital platform ( mobile app, digital weight scale, digital blood pressure monitor, biosensor with armband). Participants will have access to the community health worker and the digital platform throughout the 30-day study interval.
  Interventions: Other: Digitally-enabled CHW Care
- Usual CHW Care (Active Comparator): Patients identified by the MGH readmission database and the EHR as eligible for the study will be enrolled. Participants will be paired with a community health worker. Participants will have access to the community health worker throughout the 30-day study interval.
  Interventions: Behavioral: Usual CHW Care

INTERVENTIONS:
Other: Digitally-enabled CHW Care — Patients will be paired with a CHW and be encouraged to wear the arm biosensor continuously, take blood pressure daily, respond to short symptom assessments daily or every other day, complete weekly life quality surveys, watch weekly HF educational videos and engage in digital (e.g., video visit) and phone-based, and in-person CHW interactions. Each participant will have access to the digital platform and CHW staff during their hospitalization and for the 30 days following discharge for a typical study duration of approximately 32-35 days. Participants will complete questionnaires at the time of enrollment and at study end. Participants will also complete exit interviews in-person or via phone after the study ends.
  Arms: Intervention
Behavioral: Usual CHW Care — Patients will be paired with a CHW for 30-days. Participants will complete questionnaires at the time of enrollment and at study end. Participants will also complete exit interviews in-person or via phone after the study ends.
  Arms: Usual CHW Care

SUMMARY:
The purpose of this study is to assess the acceptability, feasibility, and preliminary effectiveness of implementing a 30-day digitally-enabled community health worker intervention compared to usual care with a community health worker in reducing heart failure 30-day readmissions within a pilot randomized controlled trial.

DETAILED DESCRIPTION:
Heart failure (HF) is a highly prevalent disease in the United States, with elevated morbidity and mortality. Nearly 6.2 million people in the US are affected by HF and this number is expected to rise to 8.5 million by 2030. Total direct medical costs of HF, mostly generated by inpatient hospitalizations, are estimated to increase from $21 billion in 2012 to $53 billion by 2030. HF is the leading cause of 30-day readmissions in the US; a quarter of these are considered to be preventable. Most patients with HF are readmitted to hospital medicine services for non-HF co-morbidities (e.g. pneumonia) with clinical, social, and behavioral factors driving readmissions. Despite numerous interventions designed to prevent readmissions, including telemetry monitoring, only marginal HF outcome improvement has been observed. HF readmission rates remain elevated and could be prevented by a multidisciplinary approach promoting better connections to and communication with clinical care teams while addressing social and behavioral barriers to HF care.

One approach that has demonstrated improved chronic disease outcomes by addressing social, behavioral, and basic clinical barriers to care- and has yet to be formally studied in HF populations- is community health workers (CHWs). CHWs are members of clinical teams who address social, economic, educational, behavioral, and basic clinical factors influencing health outcomes while fostering patient connections to care teams. CHW care delivery is one of a few interventions shown to reduce readmissions in patients with chronic disease. CHWs have basic clinical knowledge of specific conditions, along with a skillset designed to address social and behavioral drivers of health outcomes like 30-day readmissions. However, CHW care is challenged by key factors, including intensive 1:1 care delivery, limiting its scale and efficiency.

In 2016, a biotechnology company launched a HF digital platform within a mobile phone application to help reduce 30-day readmissions in patients with HF by 1) leveraging artificial intelligence to minimize false alarms in biometric monitoring, 2) promoting early identification of decline in HF patients, and 3) encouraging digital and in-person communication between patients and care teams. In preliminary findings, digital platform clinical trial data has shown promise in reducing HF 30-day readmissions. This study will investigate the effectiveness of this platform in combination with CHW care in reducing readmissions for medically and socially complex patients with HF. Through a partnership with the digital platform creators, our team has helped develop a prototype for patients with HF cared for by CHWs ("digitally-enabled" CHW care). Specifically, the aim of this proposal are to assess the acceptability, feasibility, and preliminary effectiveness of implementing a digitally-enabled CHW intervention compared to CHW care to reduce HF 30-day readmissions within a pilot RCT (n=50) My central hypothesis is that pairing patients with a digitally-enabled CHW intervention that addresses social and behavioral barriers to HF care, promotes communication with clinical care teams, and improves CHW efficiency will reduce 30-day readmissions while improving patient engagement with HF care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* HF diagnosis
* English proficiency
* Residence within 30 miles of MGH
* Being cared for by a cardiologist or primary care provider who manages their HF
* Current use and ownership of a smart phone

Exclusion Criteria:

* Cognitive deficits that prevent digital or human engagement
* Lack of health insurance
* Invoked health proxy or guardianship status
* History of smart phone use

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn Carter, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The data can be available by request only after academic journal publication. Any formal requests should be sent by external research teams and will be reviewed by the corresponding author.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available upon request after academic journal publication.
Access Criteria: Access criteria will be determined and confirmed by the corresponding author upon review of the formal data request.

REFERENCES:
- [Background] Heidenreich PA, Albert NM, Allen LA, Bluemke DA, Butler J, Fonarow GC, Ikonomidis JS, Khavjou O, Konstam MA, Maddox TM, Nichol G, Pham M, Pina IL, Trogdon JG; American Heart Association Advocacy Coordinating Committee; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Cardiovascular Radiology and Intervention; Council on Clinical Cardiology; Council on Epidemiology and Prevention; Stroke Council. Forecasting the impact of heart failure in the United States: a policy statement from the American Heart Association. Circ Heart Fail. 2013 May;6(3):606-19. doi: 10.1161/HHF.0b013e318291329a. Epub 2013 Apr 24. PMID 23616602
- [Background] McHugh MD, Ma C. Hospital nursing and 30-day readmissions among Medicare patients with heart failure, acute myocardial infarction, and pneumonia. Med Care. 2013 Jan;51(1):52-9. doi: 10.1097/MLR.0b013e3182763284. PMID 23151591
- [Background] Abdel-All M, Putica B, Praveen D, Abimbola S, Joshi R. Effectiveness of community health worker training programmes for cardiovascular disease management in low-income and middle-income countries: a systematic review. BMJ Open. 2017 Nov 3;7(11):e015529. doi: 10.1136/bmjopen-2016-015529. PMID 29101131
- [Background] Spencer MS, Kieffer EC, Sinco B, Piatt G, Palmisano G, Hawkins J, Lebron A, Espitia N, Tang T, Funnell M, Heisler M. Outcomes at 18 Months From a Community Health Worker and Peer Leader Diabetes Self-Management Program for Latino Adults. Diabetes Care. 2018 Jul;41(7):1414-1422. doi: 10.2337/dc17-0978. Epub 2018 Apr 27. PMID 29703724
- [Derived] Carter JAC, Swack N, Isselbacher E, Donelan K, Thorndike A. Feasibility, Acceptability, and Preliminary Effectiveness of a Combined Digital Platform and Community Health Worker Intervention for Patients With Heart Failure: Pilot Randomized Controlled Trial. JMIR Cardio. 2024 Aug 8;8:e59948. doi: 10.2196/59948. PMID 38959294
- [Derived] Carter J, Swack N, Isselbacher E, Donelan K, Thorndike A. Feasibility, Acceptability, and Preliminary Effectiveness of a Combined Digital Platform and Community Health Worker Intervention for Patients With Heart Failure: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Feb 6;13:e55687. doi: 10.2196/55687. PMID 38216543

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Usual CHW Care
Started | 25 | 31
Completed | 20 | 27
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual CHW Care | Total
Number analyzed (Participants) | 25 | 31 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 21 | 38
  >=65 years | 8 | 10 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] — Specific chronological age for all participants
  years | 61.6 (16.3) | 69.4 (10.3) | 65.1 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Specific gendered information for all participants
  Participants
    Female | 11 | 17 | 28
    Male | 14 | 14 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Includes multiple racial and ethnic descriptors of study participants
  Participants
    Asian, non-Hispanic | 2 | 1 | 3
    Black, non-Hispanic | 3 | 6 | 9
    Hispanic/ Latin | 2 | 2 | 4
    White, non-Hispanic | 17 | 22 | 39
    More than one race | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 25 | 31 | 56

OUTCOME MEASURES:

1. Primary Outcome: Intervention Acceptability
Description: Proportion of patients indicating that they would be willing to use the intervention again
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual CHW Care
Number analyzed (Participants) | 19 | 28
Participants | 19 | 25

2. Primary Outcome: Intervention Feasibility
Description: Proportion of patients that used the intervention during the study period
Time Frame: 30 days
Population: Given the specificity of the heart failure intervention, feasibility or use of the intervention may reflect 100% of participants being engaged with the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual CHW Care
Number analyzed (Participants) | 19 | 28
Participants | 19 | 28

3. Secondary Outcome: 30-day Readmission Rate
Description: Proportion of patients readmitted to the hospital within 30-days after hospital discharge
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual CHW Care
Number analyzed (Participants) | 19 | 28
Participants | 3 | 8

4. Secondary Outcome: 30-day Missed Appointment Rate
Description: Proportion of patients missing PCP or specialty appointments within 30-days after hospital discharge
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual CHW Care
Number analyzed (Participants) | 19 | 28
Participants | 0 | 3

5. Secondary Outcome: 30-day Emergency Department Visit Rate
Description: Proportion of patients returning to the Emergency Department within 30-days of hospital discharge
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual CHW Care
Number analyzed (Participants) | 19 | 28
Participants | 8 | 7

6. Secondary Outcome: Heart Failure Knowledge (Associated With a Subset of Participants Assessed for This Measure Prior to Being Randomized to the Intervention or Control Arm)
Description: Proportion of patients perceiving their heart failure knowledge as very good or good (per an internally validated knowledge questionnaire; very good, good, fair, poor)
Time Frame: Baseline
Population: Aim 1
Measure: Count of Participants; unit: Participants
Groups:
- Qualitative Interviews: Patients identified by the MGH readmission database and the EHR as eligible for the study will be enrolled and complete a qualitative interview via phone.
Arm/Group | Qualitative Interviews
Number analyzed (Participants) | 27
Participants | 25

7. Other Pre Specified Outcome: Patient Satisfaction
Description: Proportion of patients indicating after intervention that they were "satisfied" on a scale ranging from "satisfied" to "neutral" to "not satisfied
Time Frame: 30 days
Population: Participants indicating after intervention that they were "satisfied" on a scale ranging from "satisfied" to "neutral" to "not satisfied"
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual CHW Care
Number analyzed (Participants) | 19 | 28
Participants | 19 | 26

8. Other Pre Specified Outcome: Medication Compliance
Description: Proportion of patients demonstrating improved medication compliance on the MMAS after the intervention
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual CHW Care
Number analyzed (Participants) | 19 | 28
Participants | 8 | 5

9. Other Pre Specified Outcome: Quality of Life (Patient Perceptions and Attitudes, Functionality and Mobility)
Description: Proportion of patients demonstrating improved perceived quality of life on the KCCQ after the intervention
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual CHW Care
Number analyzed (Participants) | 19 | 28
Participants | 16 | 15

ADVERSE EVENTS:
Time Frame: 1 month
Description: By Treatment Group
  • Control- 1 (death; unrelated)
Arm/Group | Intervention | Usual CHW Care
All-Cause Mortality (participants affected / at risk) | 0/25 | 1/31
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/31
Other Adverse Events (participants affected / at risk) | 0/25 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=25) | Usual CHW Care (N=31)
Death (Cardiac disorders) | 0 (0) | 1 (1) — Fatal Cardiac Arrhythmia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT05130008/Prot_SAP_000.pdf